CLINICAL TRIAL: NCT05145036
Title: The Effect of Tai Chi Exercise Among Elders With Sarcopenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: CMUH110-REC2-107
Record Dates: First submitted 2021-10-14; First posted 2021-12-06 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Sarcopenia in Elderly; Tai Chi
MeSH Terms: interventions — Tai Ji; IPS e.max Press; Plyometric Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi exercise (Active Comparator): In addition to standard of care participants will be asked to apply Tai Chi. There are 8 movements. Each session consisted of 10 minutes of warm-up, 40 minutes of Tai Chi, and 10 minutes of cool down. The 8 movements are: Ward-off, Rollback, Push, Press, Grab, Split, Elbow strike, and shoulder strike.
  Interventions: Behavioral: Tai-Chi
- Comprehensive training (Active Comparator): In addition to standard of care participants will be asked to apply Comprehensive training. There are 3 exercises. Each session consisted of 10 minutes of warm-up, 40 minutes of Tai Chi, and 10 minutes of cool down. The 8 movements are: stretch exercise, strengthening exercise, and balance exercise.
  Interventions: Behavioral: Comprehensive training

INTERVENTIONS:
Behavioral: Tai-Chi — Tai Chi exercise could improve muscle performance, balance and have the benefit for fall down prevention in the elders and patients with frailty.
  Other Names: Ward-off; Rollback; Push; Press; Grab; Split; Elbow Strike; Shoulder Strike
  Arms: Tai Chi exercise
Behavioral: Comprehensive training — There are 3 exercises. Each session consisted of 10 minutes of warm-up, 40 minutes of Tai Chi, and 10 minutes of cool down.
  Other Names: Stretch exercise; Strengthening exercise; Balance training
  Arms: Comprehensive training

SUMMARY:
Sarcopenia has been defined as a disease which presented as low muscles strength, low muscle quantity or quality and low physical activity. The prevalence of sarcopenia is increasing with the age and it is also included in one of geriatric syndromes. Several criteria have been mentioned for diagnosis of sarcopenia, such as European Working Group on Sarcopenia in Older People (EWGSOP)、Foundation for the National Institutes of Health Biomarkers Consortium Sarcopenia Project (FNIH) and Asian Working Group for Sarcopenia (AWGS).

In European, the prevalence rate of sarcopenia is 9.25-18%; 5-7% Canadian and 14.4% Taiwanese elders have been diagnosed as sarcopenia, respectively. The sarcopenia has been found its relationship with adverse outcomes of fall down, fracture, disability, and death. The cytokines and decline in anabolic hormones play a role in the pathogenesis of sarcopenia. Tai Chi exercise is one of Qigong and well-popular in Chinese population, and is helpful to integration of body movements. Tai Chi exercise is less complicated and emphasized people's awareness of self-care which presented the relationship between human and nature. Tai Chi exercise could improve muscle performance, balance and have the benefit for fall down prevention in the elders and patients with frailty. Furthermore, Tai Chi has been found that it also could improve the muscle power and power strength in sarcopenic elders by team training. Furthermore, immune makers of inflammation process have been noted their diminishments by Qigong intervention.

The aim of this study is to investigate the effect of Tai Chi exercise in sarcopenic elders through practicing at home. The differences of muscles strength, muscle quantity or quality and physical activity after interventions would be recorded and analyzed. The cytokines related to the sarcopenia process would also be sampled.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older;
* With a diagnosis of sarcopenia [defined as EWGSOP-2] (6);
* Without planned exercise program or unplanned admission in 6 months;
* Could tolerate tests of muscle power and strength.

Exclusion Criteria:

* Uncontrolled diabetes mellitus;
* Uncontrolled cardiovascular diseases;
* Uncontrolled hypertension;
* Knee or hip prosthesis, pacemaker, fracture in the previous 6 months,
* Critical cognitive (MMSE<23)
* Mini Nutritional Assessment (MNA <17)
* Physical dysfunctions that could not tolerate our tests

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Appendicular skeletal muscle mass in kilograms | baseline
  The appendicular skeletal muscle mass is evaluated by bioelectrical impedance (BIA) analysis
Change from baseline appendicular skeletal muscle mass at 8 weeks | 8 weeks
  The appendicular skeletal muscle mass is evaluated by bioelectrical impedance (BIA) analysis
Hand grip in kilograms | baseline
  The muscle strength is evaluated with the hand-grip strength (kg) by dynamometer
Hand grip in kilograms | 8 weeks
  The muscle strength is evaluated with the hand-grip strength (kg) by dynamometer
Times Chair-stand test (5-CST) in minutes | baseline
  The 5CST is evaluated by recording the total time that patient repeat 5 times stand and sit motion from chair
Times Chair-stand test (5-CST) in minutes | 8 weeks
  The 5CST is evaluated by recording the total time that patient repeat 5 times stand and sit motion from chair

CONTACTS AND LOCATIONS:
Overall Officials: China Medicine University China Medicine University, Study Chair — China Medicine University
Locations (1):
- China Medical University Hospital, Taichung, Taiwan